CLINICAL TRIAL: NCT05843318
Title: Water Intake and Weight Control in Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Brenda Davy, Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 22-624
Record Dates: First submitted 2023-04-12; First posted 2023-05-06 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-06

CONDITIONS: Overweight and Obesity
MeSH Terms: conditions — Overweight; Obesity | interventions — Drinking

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pre-meal water + Hypocaloric diet (Experimental): premeal water ( 500 ml) before each main meal, three times per day + hypocaloric diet
  Interventions: Behavioral: Water intake and weight control in older adults - Premeal Water + hypocaloric diet
- Daily water + Hypocaloric diet (Experimental): total daily water prescription (1500 ml/d) + hypocaloric diet
  Interventions: Behavioral: Water intake and weight control in older adults - Total Daily Water + hypocaloric diet
- Hypocaloric Diet alone (Active Comparator): hypocaloric diet with not instructions regarding water intake
  Interventions: Behavioral: Water Intake and weight control in older adults - hypocaloric diet alone

INTERVENTIONS:
Behavioral: Water intake and weight control in older adults - Premeal Water + hypocaloric diet — Individuals will be randomly assigned to one of three groups. All individuals will receive counseling in a structured hypocaloric meal plan (1200-1500 kcal) that is consistent with a healthy dietary pattern as described by the Dietary Guidelines for Americans. This group will receive specific instructions for daily water intake timing and volume.
  Arms: Pre-meal water + Hypocaloric diet
Behavioral: Water intake and weight control in older adults - Total Daily Water + hypocaloric diet — Individuals will be randomly assigned to one of three groups. All individuals will receive counseling in a structured hypocaloric meal plan (1200-1500 kcal) that is consistent with a healthy dietary pattern as described by the Dietary Guidelines for Americans. This group will receive specific instructions for total daily water intake.
  Arms: Daily water + Hypocaloric diet
Behavioral: Water Intake and weight control in older adults - hypocaloric diet alone — Individuals will be randomly assigned to one of three groups. All individuals will receive counseling in a structured hypocaloric meal plan (1200-1500 kcal) that is consistent with a healthy dietary pattern as described by the Dietary Guidelines for Americans. This group will receive instructions in the hypocaloric diet, without specific fluid intake recommendations.
  Arms: Hypocaloric Diet alone

SUMMARY:
This study is a randomized controlled intervention trial in adults aged 50+ years with overweight or obesity, which will compare three groups with different diet prescriptions: 1) pre-meal water consumption (500 ml, before each main meal) with a hypocaloric diet; 2) 1500 ml water consumed throughout the day with a hypocaloric diet; 3) hypocaloric diet with no instructions regarding water consumption. Smart water bottles will objectively assess water intake timing and volume. Urine osmolality, urine volume, and serum osmolality will be used as objective indicators of compliance with the water intake prescription. We will investigate changes in perceived hunger and fullness and appetite-regulating hormones as potential mechanisms by which premeal water could improve appetite regulation. We will also investigate the impact of water consumption and hydration on executive function capabilities, which may influence intervention adherence. Although increasing water intake could be an effective weight management strategy, no evidence-based recommendations exist for the timing of water intake needed for this benefit.

ELIGIBILITY:
Inclusion Criteria:

* aged 50+ years
* BMI ≥25 kg/m2
* weight stable (+/- 2 kg) in past 6 months
* willing to provide consent and comply with study protocol

Exclusion Criteria:

* usual plain drinking water intake >1500 ml/d
* uncontrolled hypertension (>159/99 mmHg)
* medical condition requiring specialized diet prescription (eg, T2D, CHF wih fluid restriction)
* medical condition that precludes participating in a physical activity program (eg, orthopedic injury)
* current or history of GI disease (eg, Crohn's), GI surgery, or medications which impact GI function
* allergies or aversions to foods included in the test meals

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 375 (Estimated)
Dates: Start 2023-11-13 (Actual); Primary Completion 2027-12-20 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Body weight change | weeks 0 to 12 in the weight loss phase, month 0 to 12 post weight loss phase
  Body weight change in weight loss and weight loss maintenance phases

SECONDARY OUTCOMES:
Change in appetite sensations | weeks 0 to 12 in the weight loss phase, month 0 to 12 post weight loss phase
  Changes in hunger and fullness, assessed using 100mm Visual Analog Scales (VAS), in weight loss and weight loss maintenance phases. These changes may mediate adherence to the hypocaloric diet and weight loss outcomes.
Change in hydration status | weeks 0 to 12 in the weight loss phase, month 0 to 12 post weight loss phase
  Changes in hydration status, assessed using urine and serum osmolality, urine specific gravity, and serum sodium, in weight loss and weight loss maintenance phases. These changes may mediate intervention adherence.
Change in executive function (EF) | weeks 0 to 12 in the weight loss phase, month 0 to 12 post weight loss phase
  Changes in EF (attention, inhibition) assessed using ePRIME computerized tasks, in weight loss and weight loss maintenance phases. These changes may mediate intervention adherence.

OTHER OUTCOMES:
Changes in appetite hormones | weeks 0 to 12 in the weight loss phase, month 0 to 12 post weight loss phase
  Changes in appetite hormones, specifically blood concentrations of ghrelin, PYY 3-36, leptin, and CCK in response to a standardized test meal with an energy content of 25% estimated energy requirements.

CONTACTS AND LOCATIONS:
Overall Officials: Brenda Davy, PhD RDN, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Virginia Tech, Blacksburg, Virginia, United States